CLINICAL TRIAL: NCT01411878
Title: Creating Healthy Adolescents Through Meaningful Prevention Services
Brief Title: Louisville Teen Pregnancy Prevention Project
Acronym: CHAMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anita Barbee, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TP2AH000010-01-00
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Pregnancy; Sexually Transmitted Diseases
Keywords: Teen Pregnancy Prevention
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reducing the Risk (Experimental): Students will be randomly assigned to participate in Reducing the Risk training
  Interventions: Behavioral: Reducing the Risk
- Love Notes (Experimental): The second healthy relationships program for high-risk youth, Love Notes, was developed to educate participants about healthy relationships, including issues of decision-making, communication and conflict resolution, and overall safety, including the prevention of pregnancy and sexually transmitted disease (Pearson, 2009). Love Notes is a derivative of the Prevention and Relationship Enhancement Program (PREP; Stanley, Markman, & Jenkins, 2009), which is relationship marriage education program listed as an evidence-based practice (EBP) by SAMSHA (www.samhsa.gov).
  Interventions: Behavioral: Love Notes

INTERVENTIONS:
Behavioral: Reducing the Risk — Reducing the Risk: Building Skills to Prevent Pregnancy, STD and HIV (RtR) was developed by Richard Barth, MSW, Ph.D. in California. The training manual is in its 5th Edition and was last published in 2011. This curriculum is one of the first that was evaluated using an experimental design, with a longitudinal follow up (6 months and 18 months) and tested on a large group of high school students (N = 758). It is also one of the first programs to show an impact on beliefs of adolescent sexual behavior prevalence and actual behavior as well as increasing parent-child communication about abstinence and contraception (Kirby, Barth, Leland, and Fetro, 1991).
  Other Names: Comprehensive Sex Ed
  Arms: Reducing the Risk
Behavioral: Love Notes — The second healthy relationships program for high-risk youth, Love Notes, was developed to educate participants about healthy relationships, including issues of decision-making, communication and conflict resolution, and overall safety, including the prevention of pregnancy and sexually transmitted disease (Pearson, 2009). Love Notes is a derivative of the Prevention and Relationship Enhancement Program (PREP; Stanley, Markman, & Jenkins, 2009), which is relationship marriage education program listed as an evidence-based practice (EBP) by SAMSHA (www.samhsa.gov). This curriculum builds on social exchange theory and meets the needs of youth who are alienated and in need of loving personal relationships.
  Other Names: Relationship Ed
  Arms: Love Notes

SUMMARY:
This study is comparing the impact of two teen pregnancy prevention interventions, Reducing the Risk and Love Note with a non-related training on community building to determine which is most effective for which participants in delaying sexual initiation, enhancing use of condoms and other forms of birth control, decreasing sexually transmitted diseases and decreasing the number of pregnancies. The participants were 1450 youth between the ages of 14 and 19 including those from poor urban settings, those from immigrant and refugee families and those from the foster care system. Both girls and boys were be in the study. The investigators predict that girls, immigrants and refugees and foster youth will have better outcomes when participating in Love Notes, a program focused on healthy relationship formation and maintenance as a frame for how to manage the sexual aspect of relationships while boys and urban youth will have better outcomes when participating in Reducing the Risk. Both groups will have better outcomes than those in the control condition.

DETAILED DESCRIPTION:
The purpose of this research is to conduct a randomized controlled trial with three groups to test the effectiveness of various interventions aimed at reducing risky behavior by teenagers. Two intervention groups will each receive a training intervention to reduce the chances of teen pregnancy, contraction of STIs, and abusive relationships among high risk youth in the Louisville community. The wait-list control group will receive training on the unrelated topic of community building at the same time. According to the Centers for Disease Control (CDC) Youth Risk Behavior Surveillance System (YRBSS), 50% of Kentucky high school students have participated in sexual intercourse, 37% report currently being sexually active, and 14% have reported having sexual intercourse with four or more sexual partners. Furthermore, only 41% of sexually active students reported using a condom the last time they had sex. These are risky sexual practices that may lead to HIV/STI infection, as well as unintended pregnancy, within the adolescent population. Understanding the pregnancy intentions of these adolescents is not only important with regards to adolescent pregnancy, but it is also important in light of HIV and STI infection when 6% of adolescents and young adults (<20 years of age) in Kentucky have been reported as HIV positive since 2009. As of January 2009, Kentucky ranked 42nd for teenage births (where 1 is best) with a teenage birth rate of 56 per 1,000 girls ages 15-19 years of age. Kentucky was only slightly above Mississippi, which ranked 50th with a teenage birth rate of 68.4 per 1,000. Kentucky's teenage birth rate is higher than the national rate which is currently 41.9 per 1,000 girls ages 15-19 years of age. The most recent Kentucky teen birth rates in 2007 show that Jefferson County (52.34 per 1,000 ages 15-19) exceeds the birth rate of the nation. To address these issues, 1450 Louisville youth were given the opportunity to participate in one of two intervention curricula: called Reducing the Risk and Love Notes, or a waiting list control condition.

ELIGIBILITY:
Inclusion Criteria:

1. Parental Informed Consent for enrollment in the CHAMPS! CAMP and accompanying research sessions,
2. Personal assent for participation in the workshop and research sessions.
3. Age 14 to 19 years old ;
4. Affiliation with youth serving organizations, or part of a current foster youth or former foster youth alumni group.

Exclusion Criteria:

1. Age 13 or younger, 20 or older;
2. Married
3. Inability to participate verbally in English;
4. Cognitive impairment that precludes the subject from giving assent or informed consent for any reason;
5. Refusal of consent to participate in the study by their parent.
6. Already pregnant or a parent, because we are attempting primary prevention.
7. Prior participation in a comparable local program, such as Love U2.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1450 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pregnancy | 2 years
  Number of girls that get pregnant. Number of girls and times boys impregnate someone.

SECONDARY OUTCOMES:
number and type of STIs contracted | 2 years
  Number of sexually transmitted infections participants contract

CONTACTS AND LOCATIONS:
Overall Officials: Anita P Barbee, Ph.D., Principal Investigator — Kent School of Social Work University of Louisville
Locations (12):
- United States (12):
  - Department for Community Based Services: Jefferson County Region, Louisville, Kentucky
  - House of Ruth, Louisville, Kentucky
  - Presbyterian Community Center, Louisville, Kentucky
  - Jewish Family and Career Services, Louisville, Kentucky
  - Gate of Hope Ministries, Louisville, Kentucky
  - St George Community Center, Louisville, Kentucky
  - Neighborhood House, Louisville, Kentucky
  - One Plus One Equals You, Louisville, Kentucky
  - Americana Community Center, Louisville, Kentucky
  - Canaan Community Development Corporation, Louisville, Kentucky
  - Maryhurst, Louisville, Kentucky
  - The Steward's Staff, Louisville, Kentucky

REFERENCES:
- [Result] Barbee AP, Cunningham MR, van Zyl MA, Antle BF, Langley CN. Impact of Two Adolescent Pregnancy Prevention Interventions on Risky Sexual Behavior: A Three-Arm Cluster Randomized Control Trial. Am J Public Health. 2016 Sep;106(S1):S85-S90. doi: 10.2105/AJPH.2016.303429. PMID 27689500